CLINICAL TRIAL: NCT01507532
Title: Pharmacokinetic Assessment of Ceftazidime in Intermittent Hemodialysis Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: did not enroll a patient
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Marc Scheetz, Associate Professor, Midwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU00056702
Record Dates: First submitted 2012-01-03; First posted 2012-01-11 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Ceftazidime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftazidime (Other): pharmacokinetic monitoring
  Interventions: Other: pharmacokinetic monitoring

INTERVENTIONS:
Other: pharmacokinetic monitoring — pharmacokinetic monitoring
  Other Names: Fortaz

SUMMARY:
Ceftazidime is a broad spectrum cephalosporin with high activity against a variety of Gram-negative pathogens, including Pseudomonas aeruginosa. An open-label study of intravenous ceftazidime pharmacokinetics will be performed in patients undergoing intermittent hemodialysis at Northwestern Memorial Hospital to determine the clearance of ceftazidime in high flux hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are male or female adults ≥18 years of age with an expected hospital stay of at least 48 hours, who have end-stage renal disease and been receiving intermittent hemodialysis for at least 90 days.
* Eligible patients will additionally have either central or peripheral intravenous access, and will already be prescribed ceftazidime per their primary providers.
* Written informed consent in a form approved by Northwestern Memorial Hospital, Northwestern University Institutional Review Board, and Midwestern University Institutional Review Board will be completed by the patient prior to enrollment.

Exclusion Criteria:

* Patients that only receive one dose of ceftazidime in total
* Patients with potentially altered pharmacokinetic parameters (pregnant patients, burn patients, and those that are morbidly obese (BMI ≥ 40 kg/m2).
* Not meeting inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determine clearance of ceftazidime in hemodialysis | time 0 = end of infusion) up to 72 hours
  Serial blood draws will be performed at the following times in hours (time 0 = end of infusion): the time immediately before hemodialysis, 0.5, 4, and immediately before the next dose of ceftazidime. Any extra blood from samples drawn by the primary provider per routine care during the study period will also be considered for capture if it would routinely be discarded. The blood draws for this study will occur over a period of 72 hours (i.e. until the day of the following hemodialysis session).

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Scheetz, PharmD, Principal Investigator — Midwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States